CLINICAL TRIAL: NCT02592668
Title: A Feasibility Study: Epidural Stimulation to Enable Volitional Movement After Chronic Complete Paralysis in Humans.
Brief Title: Spinal Cord Injury Epidural Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: University of California, Los Angeles (Other); Reneu Health Inc. (Other); Bel13ve in Miracles Foundation (Other); The Craig H. Neilsen Foundation (Other); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Kristin Zhao, PhD, Kristin D. Zhao, Ph.D., Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 15-000510; UL1TR000135 (NIH)
Record Dates: First submitted 2015-10-22; First posted 2015-10-30 (Estimated); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Active stimulation (Experimental): Subjects will be implanted with an epidural stimulator onto the dorsal aspect of the lumbosacral spinal cord dura mater. Patients will undergo a structured program of daily physical rehabilitation, treadmill step training, and epidural stimulation to recover motor, sensory, and autonomic function. The total estimated time for the intervention is 66 weeks.
  Interventions: Device: Epidural Stimulator

INTERVENTIONS:
Device: Epidural Stimulator — Subjects will be implanted with an epidural stimulator onto the dorsal aspect of the lumbosacral spinal cord dura mater. Patients will undergo a structured program of daily physical rehabilitation, treadmill step training, and epidural stimulation to recover motor, sensory, and autonomic function.
  Other Names: Medtronic Restore ULTRA 97712

SUMMARY:
This is a feasibility study to test the use of epidural stimulation to restore volitional function previously lost due to spinal cord injury.

Previous studies conducted in animal models, performed elsewhere and here at Mayo Clinic, have shown that direct electrical stimulation of the spinal cord increases the excitability of spared neuronal connections within the site of injury, thereby enhancing signal transmission and allowing recovery of previously lost volitional function. Recently, epidural electrical stimulation of the lumbosacral spinal cord in four individuals with spinal cord injury (SCI) has restored motor and autonomic function below the level of injury. Despite positive results, further translational research is needed to validate these findings. The goal of this proposal is to perform epidural stimulation to restore volitional function in patients with SCI. In two patients, we will implant an epidural stimulator onto the dorsal aspect of the lumbosacral spinal cord dura mater. Patients will undergo a structured program of daily physical rehabilitation, treadmill step training, and epidural stimulation to recover motor, sensory, and autonomic function.

ELIGIBILITY:
Inclusion Criteria:

* Stable medical condition without *cardiopulmonary disease or *dysautonomia that would contraindicate standing or stepping with body weight support training
* No current anti-spasticity medication regimen
* Non-progressive spinal cord injury between the vertebral levels of C7 & T10
* American Spinal Injury Association grading scale of A or B
* Sensory evoked potentials are either not present or have a bilateral delay
* Segmental reflexes remain functional below the lesion
* At least 2-years post-injury.

Exclusion Criteria:

* Pregnancy at time of enrollment
* Failure to obtain consent
* Prisoners
* Children (age less than 21)
* Any patient identified as unsuitable for this protocol by the Mayo study team
* Skeletal fracture
* Osteoporosis with Dual-energy X-ray absorptiometry (DEXA) t score ≤-3.5
* Uncontrolled urinary tract infections
* Presence or history of frequent decubitus ulcers
* Clinical depression
* Drug abuse
* Painful musculoskeletal dysfunction, unhealed fracture, contracture, pressure sore, or urinary tract infection that might interfere with stand or step training
* Current anti-spasticity medication regimen
* Voluntary motor response present in leg muscles
* Volitional control during voluntary movement attempts in leg muscles as measured by electromyography (EMG) activity
* Brain influence on spinal reflexes as measured by EMG activity
* Recordable motor evoked potential in the lower limbs with transcranial magnetic stimulation
* Implanted cardiac pacemaker
* Implanted defibrillator
* Other implanted metallic or active body worn medical electronic device such as an insulin pump
* *Cardiopulmonary disease that would result in exclusion from the study will be defined as clinically diagnosed chronic obstructive pulmonary disease, cardiac failure, and heart arrhythmia that would contraindicate sudden changes in body position such as sit-to-stand and stepping
* *Excessive and uncontrolled autonomic dysreflexia characterized by symptomatic hypotension, light headedness and hypertension, flushing and bradycardia. Additionally blood pressure monitoring will be available at all times during rehabilitation and assessment times.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-01-04 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2019-02-11 (Actual)

PRIMARY OUTCOMES:
Duration of time for which subject can sit unassisted on the edge of a mat table | Approximately 50 weeks after implantation
Assessment of volitional movement of lower limbs | Approximately 50 weeks after implantation
Subject's ability to coordinate stepping on a treadmill will be measured using biomechanical and electrophysiological analyses | Approximately 50 weeks after implantation
Duration of time for which subject can stand weight bearing with minimal assistance provided as needed. | Approximately 50 weeks after implantation

SECONDARY OUTCOMES:
Change in volitional movement restoration via NeuroRecovery scale | baseline, approximately 50 weeks after implantation
Change of bladder function, as measured by the Neurogenic Bladder Symptom Score questionnaire | baseline, approximately 50 weeks after implantation
Change in sexual function as measured by the Sexual Function Questionnaire | baseline, approximately 50 weeks after implantation
Change in body thermoregulatory capacity as measured by thermoregulatory sweat testing | baseline, approximately 50 weeks after implantation
Change in lean body mass | baseline, approximately 50 weeks after implantation
Change in bone density | baseline, approximately 50 weeks after implantation
Change in sense of wellbeing as measured by the World Health Organization Quality of Life (WHOQOL-BREF) questionnaire | baseline, approximately 50 weeks after implantation
Change in sitting balance via functional reach test | baseline, approximately 50 weeks after implantation
Change in spasticity via Ashworth spasticity test | baseline, approximately 50 weeks after implantation
Change in ability of performing basic activities of daily life via spinal cord independence measure | baseline, approximately 50 weeks after implantation
Change in total body fat | baseline, approximately 50 weeks after implantation
Change in bowel function as measured by the Neurogenic Bowel Dysfunction Score questionnaire | baseline, approximately 50 weeks after implantation

CONTACTS AND LOCATIONS:
Overall Officials: Kristin D. Zhao, Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grahn PJ, Lavrov IA, Sayenko DG, Van Straaten MG, Gill ML, Strommen JA, Calvert JS, Drubach DI, Beck LA, Linde MB, Thoreson AR, Lopez C, Mendez AA, Gad PN, Gerasimenko YP, Edgerton VR, Zhao KD, Lee KH. Enabling Task-Specific Volitional Motor Functions via Spinal Cord Neuromodulation in a Human With Paraplegia. Mayo Clin Proc. 2017 Apr;92(4):544-554. doi: 10.1016/j.mayocp.2017.02.014. PMID 28385196
- [Background] Gill ML, Grahn PJ, Calvert JS, Linde MB, Lavrov IA, Strommen JA, Beck LA, Sayenko DG, Van Straaten MG, Drubach DI, Veith DD, Thoreson AR, Lopez C, Gerasimenko YP, Edgerton VR, Lee KH, Zhao KD. Neuromodulation of lumbosacral spinal networks enables independent stepping after complete paraplegia. Nat Med. 2018 Nov;24(11):1677-1682. doi: 10.1038/s41591-018-0175-7. Epub 2018 Sep 24. PMID 30250140
- [Background] Calvert JS, Grahn PJ, Strommen JA, Lavrov IA, Beck LA, Gill ML, Linde MB, Brown DA, Van Straaten MG, Veith DD, Lopez C, Sayenko DG, Gerasimenko YP, Edgerton VR, Zhao KD, Lee KH. Electrophysiological Guidance of Epidural Electrode Array Implantation over the Human Lumbosacral Spinal Cord to Enable Motor Function after Chronic Paralysis. J Neurotrauma. 2019 May 1;36(9):1451-1460. doi: 10.1089/neu.2018.5921. Epub 2018 Dec 15. PMID 30430902
- [Derived] Gill ML, Linde MB, Hale RF, Lopez C, Fautsch KJ, Calvert JS, Veith DD, Beck LA, Garlanger KL, Sayenko DG, Lavrov IA, Thoreson AR, Grahn PJ, Zhao KD. Alterations of Spinal Epidural Stimulation-Enabled Stepping by Descending Intentional Motor Commands and Proprioceptive Inputs in Humans With Spinal Cord Injury. Front Syst Neurosci. 2021 Jan 28;14:590231. doi: 10.3389/fnsys.2020.590231. eCollection 2020. PMID 33584209
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials